CLINICAL TRIAL: NCT00309218
Title: Multicenter, Open-label, Randomized Study on Steroid-free Immunosuppression, in Comparison With Daily Steroid Therapy, in Children With Stable Renal Transplant Function Under Cyclosporine (CyA) and Mycophenolate Mofetil (MMF)
Brief Title: Steroid Withdrawal in Pediatric Renal Transplant Recipients Under Cyclosporine (CyA) and Mycophenolate Mofetil (MMF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Klinik für Kinder- und Jugendmedizin (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Dr. med. Britta Hoecker, Randomized, multicenter trial on steroid withdrawal in pediatric kidney allograft recipients under CsA and MMF, Klinik für Kinder- und Jugendmedizin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BToenshoff001
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Kidney Diseases
Keywords: Pediatric renal transplantation; Steroid withdrawal; Mycophenolate Mofetil; Cyclosporine A; Stable graft function; children; renal transplantation
MeSH Terms: conditions — Kidney Diseases | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Steroid withdrawal
  Interventions: Drug: methylprednisolone
- B (Placebo Comparator): continuos Steroid treatment
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone — withdrawal of methylprednisolone in arm A and continuous Steroid Treatment in arm B

SUMMARY:
The present study investigates the safety and efficacy of steroid withdrawal in pediatric renal transplant recipients with stable graft function under concomitant immunosuppression with cyclosporine and mycophenolate mofetil.

DETAILED DESCRIPTION:
The present protocol aims to investigate the steroid-saving potential of MMF in pediatric patients after NTx. Over a 2-year period, two treatment regimes will be compared in randomized form in patients with a stable renal transplant function in the course of 12 - 24 months after transplantation (controlled first study phase):

Branch A: CyA + MMF + withdrawal of steroids over a three-month period following randomization

Branch B: CyA + MMF + 4 mg/m² methylprednisolone (or prednisolone equivalent)/day

After two years of observation, steroids in the control group (branch B) can be withdrawn optionally in conformity with the same protocol as in branch A (uncontrolled second study phase). It is to be expected that part of the patients will decide in favour of a withdrawal of steroids. In the uncontrolled second study phase, a comparison will thus be drawn among three therapy groups over a period of another 15 months (altogether 3.5 years beginning with randomization), in order to throw some light on the medium-term effect of steroid-free immunosuppression on length growth and transplant function.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18.0 years
* Bone age of boys < 15 years, of girls < 13 years
* Patients 12-24 months after renal transplantation with stable transplant function
* First or second kidney transplant, living or cadaver kidney donation
* Triple immunosuppression with cyclosporine (CyA), MMF, and daily steroids at study entry
* Patients and parents, respectively, have given their written consent after enlightenment (informed consent)

Exclusion Criteria:

* Irreversible rejection of former transplant within 6 months
* Highly reactive (> 80%) lymphocytotoxic antibodies within 12 months prior to transplantation
* Anamnestically steroid-resistant rejection of current transplant
* More than 2 acute rejection reactions prior to study entry (i.e., in the first 12-24 months after kidney transplantation) or 1 acute rejection reaction during the last 6 months before study entry
* Glomerular filtration rate (GFR) < 40 ml/min/1.73 m² (Schwartz formula) at study entry
* Acute rejection reaction or unstable transplant function (increase of serum creatinine > 20%) during the last 6 months before study entry or histologically confirmed chronic rejection reaction
* Suspected insufficient medication compliance
* Patients receiving a basic immunosuppression other than that prescribed in this protocol
* Simultaneous therapy with growth hormone after renal transplantation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 1999-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Stimulation of length growth after 24 months (controlled study phase) and 36 months (uncontrolled study phase) | 24 months

SECONDARY OUTCOMES:
Number of patients who were deprived of steroids successfully | 24 months
Transplant survival and function after 24 (controlled) and 36 (uncontrolled) months | 24 months
Incidence and severity of steroid side effects | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Toenshoff, MD, PhD, Principal Investigator — University Children's Hospital of Heidelberg, Im Neuenheimer Feld 153, D-69120 Heidelberg, Germany
Locations (1):
- University Children's Hospital, Heidelberg, Germany